CLINICAL TRIAL: NCT00460681
Title: Phase III Study of Thymopentin in Patients After Curative Resection of Small
Brief Title: Study of Thymopentin in Patients After Curative Resection of Small Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZSH-LCI-FJ-0001
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Thymopentin; Recurrence; Resection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Thymopentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Thymopentin — subcutaneously or intramuscular inject at the dosage of 10 mg every second day (twice a week) for consecutive 3 months.

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of thymopentin on the prevention of the recurrence and metastasis of small HCC after resection.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most prevalent malignancies in China, and approximately 90% of the patients with HCC are also infected with hepatitis B virus (HBV).Chronic HBV infections are a leading cause of liver cirrhosis and hepatocellular carcinoma. Surgical resection provides a potentially curative outcome for patients who are indicated to this procedure; however, survival is far from satisfactory because of the high recurrence rate, which is approximately 38-65% during the first 5 years， even for small HCC resection , it is still as high as 43.5%，and contributed to the major cause of mortality. Several approaches have been reported to decrease the recurrence rate after curative resection of HCC, such as postoperative transcatheter arterial chemoembolization (TACE) , chemotherapy , cyclic retinoic acid , and adoptive immunotherapy . However, these approaches are either controversial or require further evaluation , a substantial need for novel treatments is required urgently.

Tumor-induced immuno-suppression leads to an imbalance within the immune system, which closely related to the HCC recurrence and metastasis after resection, and an effective response is needed to eliminate residual tumor cells after removal of the major tumor tissue by surgery. Immunomodulatory peptides, like thymopentin (TP5), may act as immunomodulatory agents in cancer chemotherapy. TP5 comprises the amino acids (Arg-Lys-Asp-Val-Tyr) and represents residues 32-36 of the nuclear protein thymopoietin (TP) . A multitude of in vivo studies have shown efficacy of TP5 treatment in the therapy of various diseases including neoplastic, immune deficiency, autoimmune, and recurrent viral diseases etc. It rectifies imbalances in the immune system without observable side effects, even at very high doses. Furthermore, TP5 is able to significantly inhibit proliferation and induce apoptosis in some type of cancer lines.

Thus TP5 can not only act as an immunomodulatory factor in cancer chemotherapy or anti-HBV therapy, but also has potential as a chemotherapeutic agent in human cancer therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients who received curative resection of HBV-related small HCC (pathologically proved, solitary tumour <5cm, or two/ tumours <5cm)
* Curative resection was defined as (1) the complete resection of all tumor nodules and the cut surface being free of cancer by histological examination; (2) no macroscopic cancerous thrombus was found in the portal vein (main trunk or two major branches), hepatic veins or bile duct, (3) no extrahepatic metastasis was found
* Evidence of a positive serum HBV profile but a negative test for anti-HCV antibody
* The major organ (heart, liver,lung and kidney) function was normal

Exclusion Criteria:

* History of cardiac disease
* Active clinically serious infection
* Known history of human immunodeficiency virus (HIV) infection
* Pregnant or breast-feeding patients
* Prior use of any systemic anti-cancer treatment for HCC, eg. Chemotherapy, immunotherapy or hormonal therapy (except that hormonal therapy for supportive care is permitted). Antiviral treatment is allowed, however interferon therapy must at least 4 weeks prior randomization
* Any condition that is unstable or which could jeopardize the safety of the patient and his / her compliance in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-02; Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | three year

SECONDARY OUTCOMES:
overall survival | three year

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, MD, Study Director — Liver Cancer Institute and Zhongshan Hospital, Fudan University, 200032, Shanghai, China.
Locations (1):
- Liver Cancer Institute and Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China